CLINICAL TRIAL: NCT01209247
Title: Emergence of Fluoroquinolone Resistance in the Commensal Flora of Patients Receiving Fluoroquinolone Treatment.
Brief Title: Emergence of Fluoroquinolone Resistance in Commensal Flora
Acronym: FQEMERG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOR09005
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: All Types of Infections
Keywords: Fluoroquinolone -resistance; Commensal flora; Emergence of resistance
MeSH Terms: interventions — Administration, Rectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient treated by fluoroquinolone (Active Comparator): patient treated by fluoroquinolone. Nasal, rectal and pharyngeal swabs
  Interventions: Other: Nasal, rectal and pharyngeal swabs
- patient not receiving FQ treatment (Placebo Comparator): reference group of patients not receiving FQ treatment, but hospitalized in the same wards at the same time
  Interventions: Other: Nasal, rectal and pharyngeal swabs

INTERVENTIONS:
Other: Nasal, rectal and pharyngeal swabs — Nasal, rectal and pharyngeal swabs were performed before, during, and one month after the end of FQ treatment.

SUMMARY:
The emergence of resistance to fluoroquinolone (FQ) is a major problem worldwide. The commensal flora is the main reservoir for antibiotic resistance. Understanding the factors (environmental, patient-related, dosis-related, drug-related…) involved in the emergence of resistance to fluoroquinolones in the commensal flora of patients treated with a FQ, may help prevent it and preserve the efficiency of these important antibiotics. Samples of rectal, nasal and pharyngeal flora will be collected from hospitalized patients before receiving a FQ, at the end of the treatment and 1 month after the end of treatment. Clinical data will be collected. The incidence and risk-factors associated with the emergence of resistance to FQ will be assessed by comparing groups with and without resistance both at the end of treatment and 1 month later.

DETAILED DESCRIPTION:
Population involved: Patients hospitalized (>1day) in one of the two participating university hospitals and receiving a treatment by a fluoroquinolone (FQ) antibiotic.

Number of centers : 2 (SAINT LOUIS and BEAUJON Hospitals, ASSISTANCE PUBLIQUE HOPITAUX DE PARIS, Paris, France).

Expected number of patients : 720

Aim : To study the incidence and risk-factors involved in the emergence of resistance to FQ in the commensal flora during and after treatment by a FQ.

Methods: Nasal, rectal and pharyngeal swabs were performed before, during, and one month after the end of FQ treatment. Microbiological analysis will focus on 3 target bacterial species: Escherichia coli from the faecal flora, alpha-haemolytic streptococci from the pharyngeal flora and non-coagulase staphylococci in the nasal flora. Patients carrying resistance at day 0 in all three flora will be excluded. The incidence and risk-factors of the emergence of resistance to FQ will be assessed at the end of treatment by FQ and 1 month after the end of treatment. Patients having resistant bacteria in their flora at the end and/or after treatment will be compared with those with no resistance.

The same swabs will be collected from a reference group of patients not receiving FQ treatment, but hospitalized in the same wards at the same time as the case patients in order to eventually detect horizontal transmission of FQ-resistant strains in the hospital ward.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation >24hours in one of the participating wards Treatment by a fluoroquinolone antibiotic.

Exclusion Criteria:

* Pregnancy or breast feeding Patients refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
emergence of fluoroquinolone-resistance | 4 months
  To know the incidence and describe risk-factors involved in the emergence of fluoroquinolone-resistance in the commensal flora of patients treated by a fluoroquinolone.

CONTACTS AND LOCATIONS:
Overall Officials: De Lastours Victoire, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- De Lastours Victoire, Paris, France

REFERENCES:
- [Result] de Lastours V, Chau F, Roy C, Larroque B, Fantin B. Emergence of quinolone resistance in the microbiota of hospitalized patients treated or not with a fluoroquinolone. J Antimicrob Chemother. 2014 Dec;69(12):3393-400. doi: 10.1093/jac/dku283. Epub 2014 Jul 24. PMID 25063781
- See also: Emergence of quinolone resistance in the microbiota of hospitalized patients treated or not with a fluoroquinolone. — http://www.ncbi.nlm.nih.gov/pubmed/25063781